CLINICAL TRIAL: NCT01188629
Title: The Personal Health Care Partner Project, Conversational IT for Better, Safer Pediatric Primary Care
Brief Title: Conversational IT for Better, Safer Pediatric Primary Care
Acronym: PHP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Bill Adams, Professor of Pediatrics, Principle Investigator, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: H-26670; R18HS017248-01 (AHRQ)
Record Dates: First submitted 2010-08-24; First posted 2010-08-25 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Preventive Care; Medication Management
Keywords: Preventive Care; Medication Management; Electronic Medical Records; Automated Telephone System
MeSH Terms: interventions — Counseling

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Safety Training (Placebo Comparator)
  Interventions: Behavioral: Safety Training
- Personal Health Partner and Counseling (PHP+C) (Experimental)
  Interventions: Behavioral: Personal Health Partner and Counseling (PHP+C)

INTERVENTIONS:
Behavioral: Safety Training — IT intervention focuses on safety in the home.
  Arms: Safety Training
Behavioral: Personal Health Partner and Counseling (PHP+C) — The PHP intervention will have three primary functional areas: 1) pre-visit assessment and counseling; 2) EHR data exchange with clinician review; and 3) post-visit follow-up, re-assessment, and counseling.
  Arms: Personal Health Partner and Counseling (PHP+C)

SUMMARY:
Interactive telephony technologies offer a potentially highly effective, patient-centered communication modality by guiding parents at home through interactive discussions that can gather information and actively reinforce recommendations and treatments. Interactive telephony systems are particularly well suited for use in vulnerable populations since access to the telephone is nearly universal, and the system does not rely on reading printed text. The investigators propose to develop and evaluate an integrated patient-centered health information system, the Personal Health Partner (PHP). The PHP will use fully automated, interactive, conversations to gather personal health data and counsel parents before scheduled visits, exchange that data with the child's primary care clinician via the electronic health record (EHR), and offer personalized follow-up assessment and counseling after visits. The information technology-based approach to be evaluated in this project will link parents and children outside the clinical setting with their primary care center and will offer comprehensive assessments AND counseling to reinforce and support parental behavior change.

DETAILED DESCRIPTION:
A large gap exists between what is recommended for effective primary care of children and what actually takes place in pediatric primary care settings, especially in the areas of preventive care. Furthermore, although medication management (safety and effectiveness) issues have emerged as an important factor for children, little is known about how medication is actually used by families at home.

With growing use of the electronic health record (EHR) come new opportunities to link patient-centered information with clinical health information systems. Linkage of these systems has the potential to inform and activate parents, provide much richer data to drive decision support at the point-of-care, and to provide ongoing support for long-term behavior change following primary care visits. The use of conversational technologies as the foundation for the project offers a number of unique advantages especially the support of lower-literacy populations and near-universal access. Systems like the Personal Health Partner (PHP) represent a model for the future of ambulatory care and the sustainable, affordable delivery of higher quality and safer care by primary care clinicians in the future.

ELIGIBILITY:
Inclusion Criteria:

* Parents of children will be enrolled in the study if they meet a set of eligibility criteria which includes:

  1. Age 0 - 11 years old
  2. A primary care patient at Boston Medical Center
  3. An English speaking child and parent.

Exclusion Criteria:

* Children will be considered ineligible for the study if they plan to move away from the Boston area in less than 3 months, or are participating in another primary care research project with content that overlaps the content within this study. Currently, there are no studies being conducted that would lead to exclusion.

Max Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 475 (Actual)
Dates: Start 2007-07; Primary Completion 2011-02 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Personal Health Partner (PHP) assessment with electronic health record (EHR) data exchange before pediatric primary care visits | 2 week -1day before doctor's appointment and 1 week after appointment
  PHP assessment with EHR data exchange before pediatric primary care visits will be associated with more comprehensive preventive and medication management assessments when compared to usual care

SECONDARY OUTCOMES:
Personal Health Partner (PHP) pre-visit counseling with post-visit reinforcement | 2 week-1day before doctor's appointment and 1 week after appointment
  PHP pre-visit counseling with post-visit reinforcement will be associated with increased preventive and medication management counseling; healthier parental behaviors; and increased parental activation when compared to parents receiving usual care.

CONTACTS AND LOCATIONS:
Overall Officials: William Adams, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Walsh KE, Bacic J, Phillips BD, Adams WG. Misuse of Pediatric Medications and Parent-Physician Communication: An Interactive Voice Response Intervention. J Patient Saf. 2021 Apr 1;17(3):e207-e213. doi: 10.1097/PTS.0000000000000375. PMID 28333698
- [Derived] Adams WG, Phillips BD, Bacic JD, Walsh KE, Shanahan CW, Paasche-Orlow MK. Automated conversation system before pediatric primary care visits: a randomized trial. Pediatrics. 2014 Sep;134(3):e691-9. doi: 10.1542/peds.2013-3759. Epub 2014 Aug 4. PMID 25092938